CLINICAL TRIAL: NCT02275650
Title: The Role of Narrowband Ultraviolet B Exposure in the Maintenance of Vitamin D Levels During Winter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: maintenance_uv
Record Dates: First submitted 2014-10-19; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Vitamin D Deficiency
Keywords: calcidiol; 25(oh)d; nbUVB; cyp27A1; cyp27B1; vitamin D
MeSH Terms: conditions — Vitamin D Deficiency; Xanthomatosis, Cerebrotendinous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nbUVB (Experimental): 2 SED dose of nbUVB will be given every other week for this intervention group.
  Interventions: Radiation: nbUVB
- control (No Intervention): No nbUVB illumination will be given for the control group.

INTERVENTIONS:
Radiation: nbUVB — 2 SED nbUVB exposure will be given every other week
  Arms: nbUVB

SUMMARY:
The investigators investigated the ability of narrowband ultraviolet B (nbUVB) treatment in the maintenance of vitamin D levels achieved during the summer in Finland. The investigators randomized 37 subjects into groups of 17 and 18 subjects. The other group received 2 standard erythema doses (SED) nbUVB exposure every other week until week 24, and serum 25(OH)D levels were measured at the onset and at weeks 6, 14, 20, 26 and 30. The control group was not illuminated and serum samples were analyzed correspondingly. Punch biopsies were taken at the onset and at week 14 for CYP27A1 and CYP27B1 enzyme expression level analyses.

DETAILED DESCRIPTION:
The investigators investigated the ability of narrowband ultraviolet B (nbUVB) treatment in the maintenance of vitamin D levels achieved during the summer in Finland. The investigators randomized 37 subjects into groups of 17 and 18 subjects. The other group received 2 standard erythema doses (SED) nbUVB exposure every other week until week 24, and serum 25(OH)D levels were measured at the onset and at weeks 6, 14, 20, 26 and 30. The control group was not illuminated and serum samples were analyzed correspondingly. 6mm punch biopsies were taken at the onset and at week 14 for CYP27A1 and CYP27B1 enzyme expression level analyses.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* Fitzpacker's skin type II-IV

Exclusion Criteria:

* age under 18
* diseases that inhibit vitamin D metabolism or absorption
* Fitzpacker's skin type I
* history of skin cancer
* vitamin D substitution 1 month before baseline or during study
* sun holidays 1 month before baseline or during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
25(OH)D level | up to 30 weeks
  Serum 25(OH)D levels were measured at the onset and at weeks 6, 14, 20, 26 and 30.

SECONDARY OUTCOMES:
CYP27A1 and CYP27B1 enzyme expression levels | up to 14 weeks
  CYP27A1 and CYP27B1 enzyme expression levels will be analysed from 6mm punch biopsies at the onset and at week 14.

CONTACTS AND LOCATIONS:
Overall Officials: Toni T Karppinen, MD, Principal Investigator — Päijät Häme Central Hospital; Erna Snellman, professor, Study Director — Tampere University Hospital
Locations (2):
- Finland (2):
  - Päijät-Häme Central Hospital, Lahdenkylä, Pirkanmaa
  - Tampere University Hospital, Tampere, Pirkanmaa